CLINICAL TRIAL: NCT03304964
Title: A Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of the MMP-12 Inhibitor FP-025 After Multiple Oral Ascending Dose Administration, and to Evaluate the Effect of Food After a Single Oral Dose Administration in Healthy Subjects
Brief Title: A Phase 1, Pharmacokinetics of the MMP-12 Inhibitor FP-025 After Multiple Oral Ascending Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: FP02C-17-001
Record Dates: First submitted 2017-09-22; First posted 2017-10-09 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: FP-025, MMP-12 inhibitor
MeSH Terms: interventions — FP-025

STUDY DESIGN:
Intervention Model Description: MAD part (Part 1) - sequential multiple ascending doses; FE part (Part 2) - crossover food effect after single dose administration
Who Masked: Participant, Investigator
Masking Description: MAD part (Part 1) - double-blind; FE part (Part 2) - open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 100 mg FP-025 (b.i.d) (Experimental)
  Interventions: Drug: FP-025 (MMP-12 inhibitor)
- 200 mg FP-025 (b.i.d.) (Experimental)
  Interventions: Drug: FP-025 (MMP-12 inhibitor)
- 400 mg FP-025 (b.i.d) (Experimental)
  Interventions: Drug: FP-025 (MMP-12 inhibitor)
- 200 mg FP-025 (single dose; fasted) (Experimental)
  Interventions: Drug: FP-025 (MMP-12 inhibitor)
- 200 mg FP-025 (single dose; fed condition) (Experimental)
  Interventions: Drug: FP-025 (MMP-12 inhibitor)

INTERVENTIONS:
Drug: FP-025 (MMP-12 inhibitor) — Treatment A: 14 oral doses of 100 mg FP-025 (n=6) or placebo (n=2) in 8 days.
  Arms: 100 mg FP-025 (b.i.d)
Drug: FP-025 (MMP-12 inhibitor) — Treatment B: 14 oral doses of 200 mg FP-025 (n=6) or placebo (n=2) in 8 days.
  Arms: 200 mg FP-025 (b.i.d.)
Drug: FP-025 (MMP-12 inhibitor) — Treatment C: 14 oral doses of 400 mg FP-025 (n=6) or placebo (n=2) in 8 days.
  Arms: 400 mg FP-025 (b.i.d)
Drug: FP-025 (MMP-12 inhibitor) — Treatment D: single oral dose of 200 mg FP-025 under fasted conditions.
  Arms: 200 mg FP-025 (single dose; fasted)
Drug: FP-025 (MMP-12 inhibitor) — Treatment E: single oral dose of 200 mg FP-025 after intake of a high-fat, high-calorie breakfast (fed condition).
  Arms: 200 mg FP-025 (single dose; fed condition)

SUMMARY:
This is a single-center, phase I study consisting of 2 parts. The first part is a multiple ascending dose (MAD) part with a randomized, double-blind, placebo-controlled design in 3 treatment groups of 8 subjects (6 active; 2 placebo). The second part is a food effect (FE) part with a randomized, open-label, 2-period, 2-way crossover, single dose design in 8 subjects.

DETAILED DESCRIPTION:
MAD part (Part 1)

After assessing eligibility during a 4-week screening period, subjects will be randomized to 1 of the 3 treatments as follows:

* Treatment A: 14 oral doses of 100 mg FP-025 (n=6) or placebo (n=2) in 8 days.
* Treatment B: 14 oral doses of 200 mg FP-025 (n=6) or placebo (n=2) in 8 days.
* Treatment C: 14 oral doses of 400 mg FP-025 (n=6) or placebo (n=2) in 8 days.

FE part (Part 2)

After assessing eligibility during a 4-week screening period, 1 treatment group of 8 subjects (8 active; 0 placebo) will be randomized to a treatment sequence (D followed by E, or E followed by D):

* Treatment D: single oral dose of 200 mg FP-025 under fasted conditions, and
* Treatment E: single oral dose of 200 mg FP-025 after intake of a high-fat, high-calorie breakfast (fed condition).

The total study planned duration for each part, Part 1 and Part 2 of the study, is approximately 6 weeks, including screening period.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following inclusion criteria:

1. Males aged ≥18 and ≤65 years or postmenopausal females aged ≥18 and ≤65 years, with a BMI ≥18 kg/m2 and ≤30 kg/m2. Female subjects must be of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy or bilateral oophorectomy; or as post-menopausal females defined as 12 months amenorrhoea and follicle stimulating hormone (FSH) levels >40 IU/L.
2. A resting pulse ≥40 bpm and ≤100 bpm at screening and on Day -1.
3. A resting systolic blood pressure of ≤150 mmHg and a resting diastolic blood pressure of ≤95 mmHg at screening and on Day -1.
4. Baseline laboratory test values within reference ranges based on the blood and urine samples taken at screening and on Day -1. Out of normal ranges values may be accepted by the Investigator, if not clinically significant.
5. The subject is, in the opinion of the Investigator, generally healthy based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
6. Male subjects must use adequate contraception, if applicable, during the study and until 3 months after completion of the study.
7. Subjects participating in the FE part of the study must be willing and able to consume the entire high-fat, high-calorie breakfast in the designated timeframe.
8. Signed Informed Consent prior to any study related procedures.
9. Ability to communicate well with the Investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

Eligible subjects must meet none of the following exclusion criteria:

1. The subject has taken prescription or non-prescription medication, herbal remedies, vitamins or minerals within 2 weeks prior to the first dose of study product (or within 5 half-lives prior to the first dose of study product for any medication ingested, whichever is longer).
2. The subject has a substance abuse-related disorder or has a history of drug, alcohol and/or substance abuse deemed significant by the investigator.
3. The subject has taken any investigational products within 60 days prior to the first dose of study product.
4. The subject has a history of severe drug allergy or hypersensitivity or food allergy.
5. The subject has a history or presence of any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (in particular diabetes or pre-diabetes), haematological, dermatological, venereal, neurological, chronic infectious or psychiatric disease or other major disorder.
6. The subject has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, which has not been in remission for at least 5 years prior to the first dose of study product.
7. The subject has a history of abdominal surgery (excluding laparoscopic cholecystectomy or uncomplicated appendectomy) or thoracic or non-peripheral vascular surgery within 6 months prior to the first dose of study product.
8. The subject has any concurrent illness that may affect the particular target or absorption, distribution, and elimination of the study product.
9. The subject has had a clinically significant illness within 4 weeks prior to the first dose of study product.
10. The subject has had surgery or trauma with significant blood loss within the last 3 months prior to the first dose of study product.
11. The subject has donated blood more than 250 mL within 2 months prior to the first dose of study product.
12. The subject has tested positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV).
13. The subject is a current smoker or uses other nicotine containing products. Ex-smokers must have ceased smoking at least 6 months prior to the first dose of study product.
14. The subject has tested positive at screening or on Day -1 for drugs of abuse or alcohol.
15. A female subject who has a positive urine pregnancy test at screening or on Day -1.
16. The subject's corrected QT interval (QTcF) (Fridericia's correction) is >450 ms as read on the printout of the ECG produced by the ECG equipment and evaluated by the Investigator at screening and on Day -1. An out-of-range or abnormal ECG may be repeated. In total, 3 ECGs should be recorded consecutively and the Investigator must evaluate the triplicate ECG. If the subject's QTcF is >450 ms on at least 2 ECGs, the subject must be excluded.
17. In general, subjects should refrain from excessive physical exercise and strenuous sports activities (endurance sports) for at least 4 days before screening and Day -1.
18. The subject is, in the opinion of the Investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.
19. Legal incapacity or limited legal capacity at screening and on Day -1.
20. Employees of the Investigator or study centre, as well as first degree family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent, AEs, SAEs and ECG abnormalities up to end-of-study (EOS). | 17 days ± 2 days
  Safety evaluation will study the adverse event (AE) profile, clinical laboratory safety tests, vital signs, and ECG monitoring
Change from baseline for vital sign, ECG parameters [(QTc = QT/RR1/3.)], and clinical laboratory test for scheduled time point up to end-of-study (EOS). | 17 days ± 2 days
  Safety evaluation will study the adverse event (AE) profile, clinical laboratory safety tests, vital signs, and ECG monitoring. The ECG parameter QTc will be calculated according to Fridericia's correction using the ECG parameters QT interval (QT) and RR recorded. QTc (msec) = QT (msec)/RR (sec)1/3. QT msec will be calculated with RR sec to arrive at one reported value for QTc.

SECONDARY OUTCOMES:
Analysis of the plasma concentration-time on Day 1 (Cmax) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 1 (Tmax) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 1 (AUC0-12) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 1 (AUC0-24) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 1 (AUC0-inf) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (AI) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (Cmax) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (Tmax ) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (Cmin) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (AUC0-12) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (AUC0-inf) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (Cavg) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (FI) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (t½) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (Vss/F) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time on Day 8 (Vz/ F) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Plasma concentration-time ratio for AUC0-12 (Day 8)/AUC0-12 (Day 1) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Plasma concentration-time ratio for ratio of AUC0-12(Day 8)/AUC0-inf (Day 1) | 17 days ± 2 days
  Pharmacokinetics (PK) analysis to measure the plasma concentration of FP-025 after multiple oral ascending doses of FP-025 in healthy subjects.
Analysis of the plasma concentration-time for Cmax | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for Tmax | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for AUC0-t | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for AUC0-inf | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for Kel | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for t½ | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for CL/F | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.
Analysis of the plasma concentration-time for Vz/F | 17 days ± 2 days
  Effect of food on the Pharmacokinetics (PK) analysis after single dose administration of FP-025.

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Netherlands B.V., Petrus Campersingel 123, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abd-Elaziz K, Voors-Pette C, Wang KL, Pan S, Lee Y, Mao J, Li Y, Chien B, Lau D, Diamant Z. First-in-Man Safety, Tolerability, and Pharmacokinetics of a Novel and Highly Selective Inhibitor of Matrix Metalloproteinase-12, FP-025: Results from Two Randomized Studies in Healthy Subjects. Clin Drug Investig. 2021 Jan;41(1):65-76. doi: 10.1007/s40261-020-00981-9. Epub 2020 Dec 17. PMID 33331980